CLINICAL TRIAL: NCT03903354
Title: Relationship Between Severe Intraoperative Hyperglycemia and Infections Within 7 Days After Orthopedic Surgery
Brief Title: Intraoperative Hyperglycemia and Infections After Orthopedic Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federico Bilotta (Other)
Responsible Party: Sponsor-Investigator, Federico Bilotta, Clinical professor, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Other Study IDs: Hypergly&Infect Orth patient
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Severe Hyperglycemia; Postoperative Infection; Orthopedic Patients
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Incidence of infections within 7 days postoperatively — Measure blood glucose concentration intraoperatively and evaluate incidence of infections 7 days after surgery

SUMMARY:
Postoperative infections are a common complication. A relationship between perioperative severe hyperglycemia and postoperative infections has been found in patients undergoing craniotomy. The aim of this study is to evaluate the epidemiology of intraoperative severe hyperglycemia (BGC >180 mg/dL; 10 mmol/L) and postoperative infections (wound, urinary and prosthetic joint infection) and to investigate if severe intraoperative hyperglycemia is associated with an higher risk of early postoperative (within the 7th postoperative days) infections (wound, urinary and prosthetic joint infection).

ELIGIBILITY:
Inclusion Criteria:

* Orthopedic patients

Exclusion Criteria:

* Non-orthopedic patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We are enrolling orthopedic patients undergoing surgery.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-13 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Severe hyperglycemia and incidence of infection | Follow up of the patients for 7 days postoperatively
  Evaluate the relationship between intraoperative severe hyperglycemia and incidence of infections at 7 days follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza, Roma, RM, Italy